CLINICAL TRIAL: NCT04773379
Title: Validation of the Patient Neurotoxicity Questionnaire for Patients Suffering From Chemotherapy Induced Peripheral Neuropathy in Greek.
Brief Title: Validation of the PNQ for CIPN Patients.
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Theofilos Tsoleridis, Principal Investigator, Democritus University of Thrace
Other Study IDs: DUThrace
Record Dates: First submitted 2021-02-22; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: chemotherapy; peripheral neuropathy; questionnaire
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Patient Neurotoxicity Questionnaire (PNQ) represents a diagnostic tool concerning patients with Chemotherapy Induced Peripheral Neuropathy (CIPN). Application of such a tool in the Greek clinical praxis requires validation.

Validation consists of three stages: translation, reverse translation, and patient application. 100 oncologic patients were assessed by comparing the PNQ to the NCI-CTCAE at the chemotherapy onset and 2nd, 4th, and 6th sessions. Specific requirements of the diagnostic tool (compliance, validity, concordance, sensitivity, specificity, reliability) were statistically evaluated.

Differences between translated texts and between the reverse translation and the original were considered negligible. At the 2nd, 4th and 6th session compliance was 98%, 95% and 93% while Cronbach's α was 0,57 0,69 and 0,81 respectively. Cohen's weighted κ was 0,67 and 0,58, Spearman's ρ was 0,7 and 0,98 while AUC of the ROC was 1 and 0,9 for the sensory and the motor part respectively. The variance's linear regression analysis confirmed CIPN worsening over time (p-value<0,0001).

The Greek version remains close to the original. Compliance rates reflect easy PNQ application. Cohen's κ values highlight the physicians' tension to underestimate the patients' condition. Spearman's ρ, Cronbach's α and AUC values reflect good validity, reliability and specificity of the PNQ respectively. Finally, the linear analysis confirmed the PNQ sensitivity over time.

The PNQ validation in Greek adds a crucial tool in the physicians' armory. It can now draw the necessary information to modify the chemotherapy and analgesic treatment schemes at both preventive and acute levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 and under 80 years of age
* Patients that undergo chemotherapy for the first time
* Patients regardless of cancer type
* Patients regardless of social and education underground
* Patients able to communicate with personnel

Exclusion Criteria:

* Pediatric patients
* Preexisting neurological condition
* Patients already under chemotherapy treatment
* Patients unable to communicate with personnel

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 male or female patients from the oncology clinic of the General Hospital of Rhodes, Greece, regardless of cancer type
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in CIPN symptoms on the PNQ at the 2nd chemotherapy treatment session. | Baseline (1st chemotherapy treatment session) and up to 1 month (2nd chemotherapy treatment session).
  The PNQ is a self reported instrument assessing CIPN symptoms (sensory and motor) over time. Possible scores range from A(none) to E(severe).
Change from the 2nd chemotherapy treatment session in CIPN symptoms on the PNQ at the 4th chemotherapy treatment session. | 2nd chemotherapy treatment session and up to 2 months (4th chemotherapy treatment session).
  The PNQ is a self reported instrument assessing CIPN symptoms (sensory and motor) over time. Possible scores range from A(none) to E(severe).
Change from the 4th chemotherapy treatment session in CIPN symptoms on the PNQ at the 6th chemotherapy treatment session. | 4th chemotherapy treatment session and up to 2 months (6th chemotherapy treatment session).
  The PNQ is a self reported instrument assessing CIPN symptoms (sensory and motor) over time. Possible scores range from A(none) to E(severe).

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Rhodes, Rhodes, Dodekanese, Greece